CLINICAL TRIAL: NCT00963690
Title: CloSys Hemostatic Device U.S. Multi-Center Clinical Investigation
Brief Title: Evaluation of the CloSys Closure System as an Adjunct to Standard Compression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: CloSys Corporation (Industry)
Collaborators: Eminence Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CL-0100-01
Record Dates: First submitted 2009-08-12; First posted 2009-08-21 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Sealing the Arteriotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CloSys HD with standard compression (Experimental): CloSys Arm
  Interventions: Device: CloSys Hemostatic Device (HD); Procedure: Standard compression
- Standard compression alone (Active Comparator): Manual compression arm
  Interventions: Procedure: Standard compression

INTERVENTIONS:
Device: CloSys Hemostatic Device (HD) — Deploy CloSys HD to achieve hemostasis
  Arms: CloSys HD with standard compression
Procedure: Standard compression — Use standard compression to achieve hemostasis

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the CloSys Hemostatic Device designed to stop bleeding after an interventional procedure.

DETAILED DESCRIPTION:
To analyze the time to hemostasis (time to stop bleeding), time to ambulation (time to walk) and adverse events.

ELIGIBILITY:
General Inclusion Criteria

All answers must be YES to be eligible for the study:

1. Subject is ≥ 18 years of age;
2. Subject is willing and able to provide informed consent;
3. Subject is able to ambulate pre-procedure without difficulty;
4. Subject is able to remain supine for an extended period of time;
5. Subject is willing and able to comply with the requirements of the study protocol, including all follow-up visit evaluations;

General Exclusion Criteria

All answers must be NO to be eligible for the study:

1. Subject has a systolic blood pressure (SBP) ≥ 160 mmHg despite medical therapy;
2. Subject has a diastolic blood pressure (DBP) ≥ 100 mmHg despite medical therapy;
3. Subject has received thrombolytic therapy, such as streptokinase, urokinase, retavase, tenecteplase, or tPA, within 24 hours of the scheduled procedure;
4. Subject is lactating;
5. Subject has a life expectancy of less than one (1) year;
6. The percutaneous intervention was an emergent procedure;
7. Subject has a known coagulopathy disorder, including, but not limited to, hemophilia, sickle cell disease, or von Willebrand disease;
8. Subject has a known diagnosis of an auto-immune disease;
9. Subject has a known or suspected diagnosis of vasculitis;
10. Subject currently has an infection of any kind;
11. Subject does not have either a posterior Tibialis (PT) or dorsalis pedis (DP) pulse by doppler in ipsilateral extremity;
12. Subject has critical limb ischemia and/or severe peripheral vascular disease as identified by rest pain and/or gangrene;
13. Rutherford category five (5) or six (6);
14. Subject is currently or within the last thirty (30) days participating in another investigational drug or device study;
15. Subject is unavailable for follow-up;
16. Subject has known allergy or previous intolerance to Protamine Sulfate;
17. Subject has known allergy to shellfish;
18. Subject has had a previous closure device in the ipsilateral side within the last ninety (90) days;
19. Prior intervention or surgical procedure to the access site within the last six (6) months;
20. Subject has a planned intervention or surgical procedure prior to completion of the thirty (30) day follow-up visit;
21. Subject has received a low molecular weight (LMWH) heparin, such as, Enoxaparin sodium (Lovenox, Xaparin and Clexane) within the past twelve (12) hours;
22. Body mass index (BMI) > 45 or < 20;
23. The investigator determines the subject is otherwise not an appropriate subject for the study; 5.3.2.1 Laboratory Values Exclusion Criteria

All answers must be NO to be eligible for the study:

Within seven (7) days prior to interventional procedure or according to standard of care for percutaneous interventional procedures requiring contrast and angiography:

1. Subject is known to be, or suspected to be, pregnant (verified with a urine/blood pregnancy test);
2. Subject's pre-procedural platelet count < 100,000 103/ul;
3. Subject's hematocrit < 28%;
4. Subject's hemoglobin < 10 g/dL;
5. Subject's serum creatinine ≥ 2.5 mg/dL;
6. Prothrombin Time (PT) is not within normal limits;
7. Partial Thromboplastin Time (PTT) is not within normal limits;
8. For subjects taking warfarin (Coumadin): The subject on warfarin within 30 days has an INR ≥ 1.8 at the time of procedure;

post - Interventional Procedure Inclusion Criteria

All answers must be YES to be eligible for the study:

1. Subject has undergone a percutaneous interventional procedure utilizing a femoral arterial access;
2. Heparin is administered for anti-coagulation during the procedure;
3. Subject has an ACT ≥ 225 seconds and < 350 seconds;
4. Subject's arterial introducer sheath is 5 Fr, 6 Fr or 7 Fr;
5. Subject's arterial introducer sheath has an overall length of ≤ 15.0 cm;
6. Subject's SBP < 160 mmHg;
7. Subject's DBP < 100mmHg;
8. Subject's physical, mental, and clinical status is stable and allows for ambulation assessment four (4) hours following removal of introducer sheath; 5.3.4 Post - Interventional Procedure Exclusion Criteria

All answers must be NO to be eligible for the study:

5.3.4.1 General Exclusion Criteria

1. Subject experienced cardiogenic shock before, during, or immediately after the interventional procedure;
2. Subject has bleeding around the sheath prior to sheath removal;
3. Subject has a pseudoaneurysm before sheath removal;
4. Subject has a palpable hematoma before sheath removal;
5. Subject has evidence of a retroperitoneal bleed prior to sheath removal;
6. Subject experienced double wall punctures during vascular access;
7. Subject experienced multiple arterial punctures (> 1) during vascular access;
8. Subject has ipsilateral venous sheaths;
9. Subject had intraprocedural therapeutic thrombolysis;
10. Subject received bivalirudin(Angiomax®) before, during, or after the intervention;
11. Subject received Protamine Sulfate IV to reverse heparin received during procedure;
12. Subject has a suspected bacterial contamination of the access site;
13. Arterial access was obtained in or near a vascular graft;
14. Subject's percutaneous intervention was for the treatment of an acute myocardial infarction (MI);

Angiographic Eligibility Criteria Angiographic Inclusion Criteria

All answers must be YES to be eligible for the trial:

1. Arterial access was obtained above the femoral bifurcation;
2. Arterial access was obtained below the inguinal ligament; Angiographic Exclusion Criteria

All answers must be NO to be eligible for the trial:

1. Common femoral artery > 50% narrowing due to calcification or plaque;
2. Arteriovenous fistula present;
3. Other complication noted on femoral angiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2013-05-30 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis | 1 Hour
Time to ambulation | 6 Hours

SECONDARY OUTCOMES:
Adverse events | Within 30 days after procedure

CONTACTS AND LOCATIONS:
Overall Officials: George Adams, MD, Principal Investigator — Rex Healthcare
Locations (2):
- United States (2):
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Rex Healthcare - Rex Heart and Vascular Research, Raleigh, North Carolina